CLINICAL TRIAL: NCT00369850
Title: Investigating Bone Density and Bone Loss Without Baseline Information
Brief Title: Bone Density and Bone Loss in Postmenopausal Women With Breast Cancer Receiving Treatment in Clinical Trial IBCSG-1-98
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ETOP IBCSG Partners Foundation (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CDR0000482381; IBCSG-18-98-BS (Other: IBCSG); EU-20623 (Other: EU); IBCSG-1-98-BS (Other: IBCSG); NOVARTIS-2026703019 (Other: Novartis)
Record Dates: First submitted 2006-08-24; First posted 2006-08-29 (Estimated); Last update posted 2012-07-27 (Estimated); Status verified 2012-07

CONDITIONS: Breast Cancer; Osteoporosis
Keywords: osteoporosis; stage I breast cancer; stage II breast cancer; stage IIIA breast cancer
MeSH Terms: conditions — Breast Neoplasms; Osteoporosis | interventions — Absorptiometry, Photon

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Tamoxifen for 5 years (Experimental): Patients treated with tamoxifen for 5 years after randomisation.
  Interventions: Other: laboratory biomarker analysis; Procedure: Dual energy X-ray absorptiometry (DEXA); Procedure: Spine X-ray
- Letrozole for 5 years (Experimental): Patients treated with letrozole for 5 years after randomisation.
  Interventions: Other: laboratory biomarker analysis; Procedure: Dual energy X-ray absorptiometry (DEXA); Procedure: Spine X-ray
- Tamoxifen 2 years plus letrozole 3 years (Experimental): Patients treated with tamoxifen for 2 years and afterwards with letrozole for 3 years.
  Interventions: Other: laboratory biomarker analysis; Procedure: Dual energy X-ray absorptiometry (DEXA); Procedure: Spine X-ray
- Letrozole 2 years plus tamoxifen 3 years (Experimental): Patients treated with letrozole for 2 years and afterwards with tamoxifen for 3 years.
  Interventions: Other: laboratory biomarker analysis; Procedure: Dual energy X-ray absorptiometry (DEXA); Procedure: Spine X-ray

INTERVENTIONS:
Other: laboratory biomarker analysis — Biomarkers (C-telopeptide, osteocalcin and skeletal alkaline phosphatase) will be assessed in serum.
Procedure: Dual energy X-ray absorptiometry (DEXA) — Mone mineral density measurements of L2-L4 and hip will be performed using DEXA.
Procedure: Spine X-ray — Thoracic and lumbar X-ray (T4-L4, lateral projection) will be performed.

SUMMARY:
RATIONALE: Diagnostic procedures, such as bone mineral density testing and x-ray, help measure bone loss in women receiving treatment for breast cancer. The test results may help doctors plan better treatment.

PURPOSE: This phase III trial is studying bone density and bone loss in postmenopausal women with breast cancer receiving treatment in clinical trial IBCSG-1-98.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the effects on bone mineral density (BMD) in the L2-L4 (posterio-anterior) region of the spine and hip by assessing bone density in postmenopausal women with breast cancer receiving treatment on protocol IBCSG-1-98.
* Compare the incidence of radiological gross changes and fractures identified from spine x-rays (T4-L4) in these patients (in groups 1 and 2).
* Use longitudinal BMD measurements to estimate a linear rate of bone loss based on mixed effect models.
* Identify serum markers for bone loss to determine how they correlate with osteoporosis, microfractures, clinical fractures, and breast cancer-related bone events.

OUTLINE: This is a multicenter study and a substudy of protocol IBCSG-1-98. Patients are assigned to 1 of 3 groups according to the length of treatment they have undergone on protocol IBCSG-1-98.

* Group 1 (prior to or at the end of the second year of treatment on protocol IBCSG-1-98): Patients undergo bone mineral density (BMD) testing of the L2-L4 spine and hip at baseline and years 1, 2, 3, and 4 from baseline. They also undergo x-rays of the T4-L4 spine at baseline and years 1, 3, and 4 from baseline.
* Group 2 (after 2 years but before the end of the third year of treatment on protocol IBCSG-1-98): Patients undergo BMD testing of the L2-L4 spine and hip at baseline and years 1, 2, and 3 from baseline. They also undergo x-rays of the T4-L4 spine at baseline and years 2 and 3 from baseline.
* Group 3 (after 3 years but before the end of the fifth year of treatment on protocol IBCSG-1-98): Patients undergo BMD testing of the L2-L4 spine and hip at baseline and years 1 and 2 from baseline (for patients in 4th year of treatment) or year 1 from baseline (for patients in 5th year of treatment).

Patients undergo blood collection at baseline and periodically during study for biomarker correlative study.

PROJECTED ACCRUAL: A total of 660 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of breast cancer

  * Resected disease
* Enrolled on protocol IBCSG-1-98

  * Receiving adjuvant endocrine therapy comprising 1 of the following regimens:

    * Letrozole
    * Tamoxifen
    * Letrozole after 2 years of tamoxifen
    * Tamoxifen after 2 years of letrozole
  * Not yet completed 5 years of treatment
* No breast cancer recurrence or second primary cancer
* No known, symptomatic bone disease, including osteomalacia or osteogenesis imperfecta
* No prior registration to protocol IBCSG-1-98 Bone Mineral Density substudy
* Hormone receptor status:

  * Estrogen receptor-positive and/or progesterone receptor-positive tumor

PATIENT CHARACTERISTICS:

* Female
* Postmenopausal
* No uncontrolled thyroid or parathyroid disease, Cushing's disease, or other pituitary diseases
* No malabsorption syndrome or clinically relevant vitamin D deficiency
* No patients for whom the bone density determination is impossible

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* More than 1 year since prior and no concurrent anticonvulsants
* More than 6 weeks since prior and no concurrent corticosteroids (at doses > the equivalent of 5 mg/day prednisone) for > 2 weeks total
* No prior or concurrent sodium fluoride (at daily doses ≥ 5 mg/day) for > 1 month
* More than 12 months since prior and no concurrent anabolic steroids
* More than 6 months since prior treatment, either investigational or not, for the prevention of osteoporosis (excluding calcium or cholecalciferol [vitamin D])
* No concurrent raloxifene
* Concurrent therapeutic intervention for osteoporosis comprising bisphosphonates allowed
* Concurrent warfarin allowed provided it is given for ≤ 4 weeks

Min Age: 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 458 (Actual)
Dates: Start 2004-05; Primary Completion 2008-05 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Relative percent change of bone mineral density (BMD) form baseline to after 2, 3, 4, or 5 years of treatment on protocol IBCSG-1-98 | 5 years after randomisation to BIG 1-98
Recovery of BMD at 1 year after the completion of treatment on protocol IBCSG-1-98 | 6 years after randomisation to BIG 1-98
Proportion of patients with BMD below the absolute threshold value for osteoporosis | 5 years after randomisation to BIG 1-98
Relative percent change in markers of bone resorption from baseline to after 2, 3, 4, or 5 years of treatment on protocol IBCSG-1-98 | 5 years after randomisation to BIG 1-98
Recovery of the markers of bone resorption at 1 year after the completion of treatment on protocol IBCSG-1-98 | 6 years after randomisation to BIG 1-98

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Aebi, MD, Study Chair — Insel Gruppe AG, University Hospital Bern; Andrea Decensi, MD, Study Chair — European Institute of Oncology
Locations (16):
- Australia (2):
  - Institute of Oncology at Prince of Wales Hospital, Randwick, New South Wales
  - Royal Brisbane and Women's Hospital, Brisbane, Queensland
- Institut Bergonie, Bordeaux, France
- Italy (3):
  - Centro di Riferimento Oncologico - Aviano, Aviano
  - Ospedali Riuniti di Bergamo, Bergamo
  - European Institute of Oncology, Milan
- Dunedin Hospital, Dunedin, New Zealand
- Instituto Nacional de Enfermedades Neoplasicas, Lima, Peru
- Groote Schuur Hospital, Cape Town, South Africa
- Hospital Ruber Internacional, Madrid, Spain
- Switzerland (6):
  - Kantonspital Aarau, Aarau
  - Inselspital Bern, Bern
  - Centre Hospitalier Universitaire Vaudois, Lausanne
  - Ospedale Beata Vergine, Mendrisio
  - Kantonsspital - St. Gallen, Sankt Gallen
  - Regionalspital, Thun

REFERENCES:
- [Derived] Decensi A, Sun Z, Guerrieri-Gonzaga A, Thurlimann B, McIntosh C, Tondini C, Monnier A, Campone M, Debled M, Schonenberger A, Zaman K, Johansson H, Price KN, Gelber RD, Goldhirsch A, Coates AS, Aebi S. Bone mineral density and circulating biomarkers in the BIG 1-98 trial comparing adjuvant letrozole, tamoxifen and their sequences. Breast Cancer Res Treat. 2014 Apr;144(2):321-9. doi: 10.1007/s10549-014-2849-2. Epub 2014 Feb 1. PMID 24487691